CLINICAL TRIAL: NCT04690452
Title: Evaluation of the Efficacy and Mechanisms of Change of Compassion Cultivation Training in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Nirakara Institute (Unknown)
Responsible Party: Principal Investigator, Blanca Rojas, Assistant Professor Faculty of Medicine, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BRLUCM2020-1
Record Dates: First submitted 2020-12-22; First posted 2020-12-30 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Stress; Depression; Anxiety; Burn Out; Well-being; Resilience; MIndfulness; Compassion; Self-Compassion; Empathy
Keywords: Compassion; Medical Student; Health; Training program; CCT
MeSH Terms: conditions — Depression; Anxiety Disorders; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Medical students during academic year 2020-21 will be asked to participate in the present study. Once inclusion criteria are met, each participant will be randomly assigned to the experimental group or waitlist control. Randomization will be performed by using a computer-generated sequence
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention condition (Experimental): Intervention group that receive a standardized 8 weeks Compassion Cultivation Training from a faculty member certified CCT© instructor (https://www.compassioninstitute.com/about-us/teacher-directory/)
  Interventions: Behavioral: Compassion Cultivation Training
- Waitlist control condition (Other): The participants assigned to the waitlist control will fill in the same questionnaires as the intervention group at the different time points (i.e., pre, post, 2-month and 6-month follow-ups).
  Two months after finishing the intervention, will become participants of a CCT© program themselves given by the same faculty member certified CCT© teacher as for the experimental group.
  Interventions: Behavioral: Compassion Cultivation Training

INTERVENTIONS:
Behavioral: Compassion Cultivation Training — The Compassion Cultivation Training (CCT©) is an 8-week standardized meditation program conducted in groups of 15-20 participants and consisting of weekly 2 hour on-line sessions with 20-30 minutes of daily formal meditation practices and informal compassion practices. The CCT© program will be guided by a certified instructor form the Center for Compassion and Altruism Research and Education at Stanford University. The CCT© program comprises six sequential steps: 1) Settling the mind; 2) Loving-kindness and compassion for a loved one; 3) Self-directed loving-kindness and compassion; 4) Common humanity; 5) Cultivating compassion for others; and 6) Active compassion (Tonglen).

SUMMARY:
The aim of this randomized, waitlist controlled trial is to examine the efficacy of the Compassion Cultivation Training (CCT©) in reducing psychological distress (i.e., stress, anxiety and depression) and burnout symptoms while improving psychological well-being medical students. The second goal of the study is to examine whether mindfulness and compassion-related variables as well as emotional-cognitive emotional regulation processes mediate the psychological distress and well-being changes.

The effects of the CCT© program will be measured by means of self-report questionnaires involving different domains (mindfulness, compassion, distress, and well-being measures) at different time points (pre-intervention, inter-session assessment, post-intervention, 2-month and 6-month follow-up).

DETAILED DESCRIPTION:
Compassion and empathy are essential components of health care quality. Several studies have found a significant decrease in empathy and compassion levels during medical school and residency (Hojat, 2004; Bellini, 2005; Stephen, 2006; Neumann, 2011). However, compassion training is usually excluded from medical education. Compassion training in medical students can increase their wellness and decreased burnout (Weingartner, 2019), which in turn improves patients clinical outcomes (Kim, 2004; Rakel, 2009; Hojat, 2011; Attar 2012; Del Canale, 2012; Steinhausen, 2014; Trzeciak, 2017; Moss, 2019). Given that compassion can be trained through standardized interventions (Stephen, 2006; Hojat, 2009a; Goetz, 2010; Kelm, 2014) and educational programs (Patel, 2019), it highlight the need to investigate interventions aimed to improving both, provider self-care and patient care.

Hypothesis:

* Compassion Cultivation Training (CCT©) program would improve psychological well-being while reducing psychological distress (stress, anxiety and depression) and burnout symptoms in medical students as compared to a waitlist control group.
* These improvements would be maintained at 2 and 6 months after finishing the program.
* Mindfulness and compassion changes and emotional-cognitive emotional regulation processes would mediate the relationship between the program and the psychological distress and well-being changes.
* Compassion skills after the program will be a protective factor for stress and worry produced by COVID-19 pandemic.

Procedure:

The study will follow a randomised waitlist controlled trial with five assessment moments (i.e., pre, inter-session, post, 2-month and 6-month follow-ups). Participants will be recruited via constitutional email and the informative screens of the Medical School at Complutense University of Madrid. Participants will be randomized to either CCT© group (N=20) or waiting list control group (N=20). The procedure will include an online assessment via Qualtrics software at the different time points, as well as the completion of a "practice diary" as the inter-session assessment one per week the day before each session.

Program description:

The Compassion Cultivation Training (CCT©) is an 8-week evidence-based standardized meditation program designed at Standford University. The CCT© is aimed at cultivating compassion and empathy toward oneself and others. The program is conducted in groups of 15-20 participants and consisting of weekly 2 hour on-line sessions (due to COVID-19 restrictions) with 20-30 minutes of daily formal meditation practices and informal compassion practices. The CCT© program will be guided by a certified instructor from the Compassion Institute. Program adherence and fidelity will be monitored through revisions of the recorded sessions. The CCT© program comprises six sequential steps: 1) Settling the mind; 2) Loving-kindness and compassion for a loved one; 3) Self-directed loving-kindness and compassion; 4) Common humanity; 5) Cultivating compassion for others; and 6) Active compassion (Tonglen).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or more.
* Medical students at University Complutense of Madrid.
* Fluency in oral Spanish
* Providing written, informed consent
* Attendance commitment to all sessions of the program
* Internet and computer access

Exclusion Criteria:

* Severe mental disorder in active phase.
* Being under alcohol and other drugs influence during weekly sessions and assessments
* Participation in another meditation standardized program during CCT©.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Change in Compassion- Compassion to others at pre, post-intervention and at 2 and 6 months | up to 6 months.
  Compassion Scale Pommier (CSP; Pommier et al., 2020).
Change in Compassion- Self-compassion at pre, post-intervention and at 2 and 6 months | up to 6 months.
  Self- Compassion Scale (SCS-SF; Raes et al., 2011).
Change in Empathy at pre, post-intervention and at 2 and 6 months | up to 6 months.
  Interpersonal Reactivity Index (IRI, Davis, 1980).
Change in Psychological distress- feelings of stress, anxiety and depression at pre, post-intervention and at 2 and 6 months | up to 6 months.
  Depression Anxiety Stress Scales (DASS- 21; Lovibond, & Lovibond, 1995).
Change in General well-being at pre, post-intervention and at 2 and 6 months | up to 6 months.
  Pemberton Happiness Index (PHI, Hervas, & Vazquez, 2013).

SECONDARY OUTCOMES:
Change in Mindfulness at pre, post-intervention and at 2 and 6 months | up to 6 months.
  Five Facet Mindfulness Questionnaire (FFMQ; Baer et al., 2006).
Change in Burnout at pre, post-intervention and at 2 and 6 months | up to 6 months.
  Maslach Burnout Inventory (Maslach & Jackson, 1981)
Change in Resilience at pre, post-intervention and at 2 and 6 months | up to 6 months.
  Brief Resilience Scale (BRS; Smith et al., 2008).
Change in Emotion regulation at pre, post-intervention and at 2 and 6 months | up to 6 months.
  Difficulties in Emotion Regulation Scale (DERS, Gratz & Roemer, 2004).
Change in Adherence to the program | up to 8 weeks
  Single-item to measure daily formal meditation practices and informal compassion practices.
Changes in State measures during intervention | up to 8 weeks
  Single-item to measure state changes in: compassion, mindfulness, psychological distress, well-being, and cognitive-emotional regulation processes

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Rojas, M.D., PhD, Principal Investigator — Universidad Complutense Madrid
Locations (1):
- Universidad Complutense Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hojat M, Mangione S, Nasca TJ, Rattner S, Erdmann JB, Gonnella JS, Magee M. An empirical study of decline in empathy in medical school. Med Educ. 2004 Sep;38(9):934-41. doi: 10.1111/j.1365-2929.2004.01911.x. PMID 15327674
- [Background] Bellini LM, Shea JA. Mood change and empathy decline persist during three years of internal medicine training. Acad Med. 2005 Feb;80(2):164-7. doi: 10.1097/00001888-200502000-00013. PMID 15671323
- [Background] Stepien KA, Baernstein A. Educating for empathy. A review. J Gen Intern Med. 2006 May;21(5):524-30. doi: 10.1111/j.1525-1497.2006.00443.x. PMID 16704404
- [Background] van Donselaar CA, Habbema JD. Recurrence after first seizure. Lancet. 1991 Jan 5;337(8732):46. doi: 10.1016/0140-6736(91)93361-c. No abstract available. PMID 1670661
- [Background] Weingartner LA, Sawning S, Shaw MA, Klein JB. Compassion cultivation training promotes medical student wellness and enhanced clinical care. BMC Med Educ. 2019 May 10;19(1):139. doi: 10.1186/s12909-019-1546-6. PMID 31077192
- [Background] Kim SS, Kaplowitz S, Johnston MV. The effects of physician empathy on patient satisfaction and compliance. Eval Health Prof. 2004 Sep;27(3):237-51. doi: 10.1177/0163278704267037. PMID 15312283
- [Background] Rakel DP, Hoeft TJ, Barrett BP, Chewning BA, Craig BM, Niu M. Practitioner empathy and the duration of the common cold. Fam Med. 2009 Jul-Aug;41(7):494-501. PMID 19582635
- [Background] Hojat M, Louis DZ, Markham FW, Wender R, Rabinowitz C, Gonnella JS. Physicians' empathy and clinical outcomes for diabetic patients. Acad Med. 2011 Mar;86(3):359-64. doi: 10.1097/ACM.0b013e3182086fe1. PMID 21248604
- [Background] Attar HS, Chandramani S. Impact of physician empathy on migraine disability and migraineur compliance. Ann Indian Acad Neurol. 2012 Aug;15(Suppl 1):S89-94. doi: 10.4103/0972-2327.100025. PMID 23024571
- [Background] Del Canale S, Louis DZ, Maio V, Wang X, Rossi G, Hojat M, Gonnella JS. The relationship between physician empathy and disease complications: an empirical study of primary care physicians and their diabetic patients in Parma, Italy. Acad Med. 2012 Sep;87(9):1243-9. doi: 10.1097/ACM.0b013e3182628fbf. PMID 22836852
- [Background] Steinhausen S, Ommen O, Antoine SL, Koehler T, Pfaff H, Neugebauer E. Short- and long-term subjective medical treatment outcome of trauma surgery patients: the importance of physician empathy. Patient Prefer Adherence. 2014 Sep 18;8:1239-53. doi: 10.2147/PPA.S62925. eCollection 2014. PMID 25258518
- [Background] Moss J, Roberts MB, Shea L, Jones CW, Kilgannon H, Edmondson DE, Trzeciak S, Roberts BW. Healthcare provider compassion is associated with lower PTSD symptoms among patients with life-threatening medical emergencies: a prospective cohort study. Intensive Care Med. 2019 Jun;45(6):815-822. doi: 10.1007/s00134-019-05601-5. Epub 2019 Mar 25. PMID 30911803
- [Background] Hojat M. Ten approaches for enhancing empathy in health and human services cultures. J Health Hum Serv Adm. 2009 Spring;31(4):412-50. PMID 19385420
- [Background] Cruz A, Buhling M, Seibel K. [Double blind study of migraine therapy with etilefrine pivalate]. Arzneimittelforschung. 1985;35(7):1086-9. German. PMID 2864937
- See also: The Center for Compassion and Altruism Research and Education — http://ccare.stanford.edu/
- See also: Compassion Institute — http://www.compassioninstitute.com/
- See also: Center for Mindful Self-Compassion — http://self-compassion.org/
- See also: The Compassionate Mind Foundation — http://www.compassionatemind.co.uk